CLINICAL TRIAL: NCT03997695
Title: A Comparison of the Effects of Core Stabilization Exercise Plus Kinesio Taping to Exercise Alone on Pain, Fatigue, Health Status, Quality of Life, Sleep Quality and Depression in Woman With Fibromyalgia
Brief Title: Effects of Core Stabilization Exercise Plus Kinesio Taping in Woman With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Fibromyalgia; Exercise; Rheumatic Diseases
Keywords: Fibromyalgia; Exercise; Kinesio Taping
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stabilization exercise group (Active Comparator): Core stabilization exercise (CSE):
  The CSE program was carried out 2 days a week for 6 weeks (12 sessions) by supervisor physiotherapist. The CSE program aimed to perform neutral spine and activation of core muscles. Prior to the CSE program, participants were informed about core musculature and their function.The 6-weeks CSE program was performed in stages with gradual progression according to the stages of motor learning and sensory motor integration as static, dynamic, and functional.
  Interventions: Other: Core stabilization exercise group
- Core stabilization exercise plus kinesio taping group (Experimental): Core stabilization exercise (CSE):
  The CSE program was carried out 2 days a week for 6 weeks (12 sessions) by supervisor physiotherapist. The CSE program aimed to perform neutral spine and activation of core muscles. Prior to the CSE program, participants were informed about core musculature and their function.The 6-weeks CSE program was performed in stages with gradual progression according to the stages of motor learning and sensory motor integration as static, dynamic, and functional.
  Kinesio Taping:
  The Kinesio Taping was carried out 2 days a week for 6 weeks (12 sessions) by experienced and certificated physiotherapist. Kinesio taping was applied to spinal region.
  Interventions: Other: Core stabilization exercise plus kinesio taping group

INTERVENTIONS:
Other: Core stabilization exercise group — The CSE program was carried out 2 days a week for 6 weeks (12 sessions) by supervisor physiotherapist. The CSE program aimed to perform neutral spine and activation of core muscles. Prior to the CSE program, participants were informed about core musculature and their function.The 6-weeks CSE program was performed in stages with gradual progression according to the stages of motor learning and sensory motor integration as static, dynamic, and functional.
  Arms: Core stabilization exercise group
Other: Core stabilization exercise plus kinesio taping group — The CSE program was carried out 2 days a week for 6 weeks (12 sessions) by supervisor physiotherapist. The CSE program aimed to perform neutral spine and activation of core muscles. Prior to the CSE program, participants were informed about core musculature and their function.The 6-weeks CSE program was performed in stages with gradual progression according to the stages of motor learning and sensory motor integration as static, dynamic, and functional.
  Arms: Core stabilization exercise plus kinesio taping group

SUMMARY:
This study aimed to compare the effectiveness of a 6-week core stabilization exercise (CSE) program with and without kinesio taping on pain, fatigue, health status, quality of life, sleep quality and depression in woman with fibromyalgia.

Participants were allocated into two groups as CSE and CSE plus kinesio taping group. Pain, fatigue, health status, quality of life, sleep quality and depression were assessed at the baseline and after 6-weeks treatment.

DETAILED DESCRIPTION:
A 6-weeks prospective randomized controlled trial examined the effects of core stabilization exercise (CSE) plus kinesio taping (KT) compared to CSE alone on pain, fatigue, health status, quality of life, sleep quality and depression in woman with FM. The trial was approved by the Ethics committee of Ankara Yildirim Beyazit University (Approval time and number: 17.01.2018-14). The study was performed in compliance with Helsinki Declaration where applicable. The patient's recruitment started in February 2018. The patients diagnosed with Fibromyalgia according to the criteria of the 1990 American College of Rheumatology participated in the study. Prior to the treatment and after 6-weeks treatment, participants' pain level, fatigue, health status, quality of life (QoL), psychological status and sleep quality were assessed. Assessments were realized by face-to-face interview method.Patients who participated in CSE group performed CSE program alone, whereas patients in CSE+KT group performed CSE program with KT application. The treatment was carried out 2 days a week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Fibromyalgia, being woman, having moderate or severe pain according to Visual Analog Scale, 18-65 years of age and being volunteer for the study

Exclusion Criteria:

* having neurologic, infectious, and endocrine diseases, malignancy, being pregnant, severe psychological disorders, any changing of medications during treatment, being allergic to taping, any condition interfering with exercise (advanced cardiac, respiratory or musculoskeletal problems), and intervention including exercise program or physical therapy in the last 6 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain level | Two years
  Pain level was assessed with Visual Analog Scale.

SECONDARY OUTCOMES:
Health Status | Two years
  Health status of participants were assessed with Turkish version of Fibromyalgia Impact Questionnaire.
Life Quality | Two years
  Quality of Life was assessed with Turkish version of Nottingham Health Profile
Depression | Two years
  Depression was assessed with Turkish version of Beck Depression Inventory
Sleep Quality | Two years
  Sleep quality was assessed with Jenkins Sleep Scale.
Fatigue | Two years
  Fatigue was assessed with Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Oğuzhan Mete, PT, Study Chair — Research Assistant
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No